CLINICAL TRIAL: NCT03274427
Title: The Efficacy and Safety of TACE Combined With Arginine Hydrochloride and Trimetazidine Hydrochloride Tablets in With Hepatocellular Carcinoma. A Multicenter, Open, Randomized, Prospective Study
Brief Title: Treatment of Intermediate-stage Hepatocellular Carcinoma
Acronym: TIHCC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Collaborators: First Affiliated Hospital of Xinjiang Medical University (Other); Luoyang Central Hospital (Other); Nanyang Central Hospital (Other); Anyang Tumor Hospital (Other); Shenma Medical Group General Hospital (Other); First People's Hospital of Shangqiu (Other); Jiaozuo third people's hospital (Unknown)
Responsible Party: Principal Investigator, Zujiang YU, The director of infectious diseases department, The First Affiliated Hospital of Zhengzhou University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HETCT-002
Record Dates: First submitted 2017-08-27; First posted 2017-09-07 (Actual); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: HCC
MeSH Terms: interventions — Arginine; Trimetazidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- One-drug Regimes (Experimental): Basic drugs therapy of HCC by TACE.
  Interventions: Device: Basic drugs therapy of HCC by TACE
- Two-Drug Regimens (Experimental): Basic drugs therapy of HCC by TACE; Arginine hydrochloride
  Interventions: Device: Basic drugs therapy of HCC by TACE; Drug: Arginine hydrochloride
- Three-Drug Regimens (Experimental): Basic drugs therapy of HCC by TACE; Arginine hydrochloride;Trimetazidine hydrochloride
  Interventions: Device: Basic drugs therapy of HCC by TACE; Drug: Arginine hydrochloride; Drug: Trimetazidine hydrochloride

INTERVENTIONS:
Device: Basic drugs therapy of HCC by TACE — Basic drugs include: 1. Molecular targeted drugs for HCC：apatinib; 2. Antiviral drugs (ETV or TDF) should be given to patients who were infected with HBV or HCV; 3. Patients with liver dysfunction should be treated with conventional hepatoprotective agents drugs (including glycyrrhizin, reduced glutathione, vitamin C，etc); 4. Patients with ascites symptoms should be treated with furosemide and spironolactone according to the urine volume, and they also should be treated with proton pump inhibitors in the prevention of gastrointestinal bleeding; 5. Other basic diseases were treated routinely.
  Other Names: TACE
Drug: Arginine hydrochloride — Arginine hydrochloride injection 5g/dose; 40g/d; ivgtt; sustained medication for 24 days; drug withdrawal for 4 days.
  Other Names: AH
  Arms: Three-Drug Regimens; Two-Drug Regimens
Drug: Trimetazidine hydrochloride — Trimetazidine hydrochloride, 20mg/tablet, 40mg, twice a day.
  Other Names: TH
  Arms: Three-Drug Regimens

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of transarterial chemoembolization (TACE) combined with arginine hydrochloride and trimetazidine hydrochloride tablets in the treatment of patients with hepatocellular carcinoma.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the sixth most common cancer and the second leading cause of cancer-related deaths in the world. Because HCC is insidious and early diagnosis is difficult, most patients have locally advanced or distant metastasis at the time of diagnosis. So they are not suitable candidates for curative treatments by resection or transplantation. Currently, Sorafenib is the only choice approved by FDA for advanced HCC, although it prolongs the survival for less than 3 months. Transarterial chemoembolization (TACE) is an important method of minimally invasive therapy in the comprehensive treatment of liver cancer. As a kind of combined treatment, it can obviously prolong the survival time of the patients. Recently, metabolomics studies of HCC have shown that typical Warburg effect was observed in hepatoma carcinoma cells. Arginine hydrochloride is a new anticancer drug in the treatment of liver cancer, which is mainly aimed at the pathway of energy metabolism. Trimetazidine hydrochloride may play an anti-tumor role by inhibiting fatty acid oxidation. The investigators have been proceeding this trial to evaluate the efficacy and safety of transarterial chemoembolization (TACE) combined with arginine hydrochloride and trimetazidine hydrochloride tablets in the treatment of patients with hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* 1. Ages 18-65 years
* 2. The diagnosis of HCC: in accordance with "diagnostic and treating standards on primary liver cancer" (2011 Edition) or histological/cytological diagnosis of primary liver cancer
* 3. Un-resectable HCC who are eligible for TACE: patients with developing primary liver cancer of Barcelona stage(BCLC) B; multiple nodules (less than 5, the total diameter of less than 20 cm), no invasion, no symptoms; refusing open surgical treatment and volunteering for the treatment
* 4. There are CT or MRI measurable lesions
* 5. No major vascular invasion or extra hepatic metastasis
* 6. Child-Pugh liver function class A/B(score: ≤7)
* 7. Performance status 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) scale in one week before admission
* 8. Estimated survival time > 3 months
* 9. HBV DNA<2000 IU/ml（10^4 copies/ml); or HBV DNA≥2000 IU/ml and are accepting effective antiviral therapy
* 10. The major organ function is normal. that is meeting the following standards:

  1. Blood routine examination: (No blood transfusion, no G-CSF and no medication were corrected within 14 days before screening)

     a.HB≥80g/L； b.ANC≥1.5×109/L；c.PLT≥50×109/L；
  2. Biochemical examination: (ALB was not transfused within 14 days before screening) a.ALB ≥29 g/L； b.ALT和AST<5ULN；c.TBIL ≤3ULN；d.creatinine ≤1.5ULN( albumin and bilirubin, two indicators of Child-Pugh liver function class, can only have one for 2 points)
* 11. For women of childbearing age, the results of serum/urine pregnancy tests must be negative within 7 days before initiation of treatment. All men and women who participate in the study have to take reliable contraceptive measures within the trial and eight weeks after the trial is completed
* 12. volunteers must signed informed consent

Exclusion Criteria:

* 1. Diffuse hepatocellular carcinoma
* 2. Vascular invasion, including portal vein tumor thrombus
* 3. Extra hepatic metastasis
* 4. Decompensated Cirrhosis: Child-Pugh liver function class B/C(score: >8); jaundice; hepatic encephalopathy; refractory ascites; hepatorenal syndrome
* 5. With a history of alimentary tract hemorrhage or a definite tendency of gastrointestinal bleeding, such as varices of fundus of stomach and esophagus with bleeding risk; local active ulcer lesions; fecal occult blood ≥（++）
* 6. Contraindication of embolization: patients with severe hepatic flow or portosystemic shunt; the lesion was too large, and the majority of two lobe were occupied by the lesions
* 7. Patients whose target lesion has been treated locally: resection of hepatic carcinoma; radio frequency ablation; TACE; local treatment was taken within 4 weeks; patients who have previously been given radiotherapy, chemotherapy, or targeted drugs
* 8. Patients with hepatobiliary cell carcinoma, mixed cell carcinoma or lamellar cell carcinoma; in the past (within 5 years) or at the same time suffering from other untreated malignant tumors; excluding cured basal cell carcinoma and carcinoma in situs of cervix
* 9. Patients who are undergoing liver transplantation or have a history of organ transplantation(excluding the patient who has undergone liver transplantation before)
* 10. Patients with an allergic history of arginine hydrochloride and trimetazidine hydrochloride
* 11. The blood pressure can not be reduced to the normal range by the antihypertensive drug treatment in patients with hypertension(systolic pressure>140 mmHg, diastolic pressure>90 mmHg)
* 12. Patients with myocardial ischemia or myocardial infarction over grade II or a poorly controlled arrhythmia (including QTc interval: men ≥ 450 ms; women ≥ 470 ms)
* 13. Cardiac functional insufficiency of grade III to IV according to NYHA standard; echocardiography: LVEF<50%
* 14. Many factors that influence oral medication, such as unable to swallow; chronic diarrhea; intestinal obstruction; the situations which significantly affect the use and absorption of drugs
* 15. Abdominal fistula, gastrointestinal perforation, or abdominal abscess occurred within 28 days before participating the study
* 16. Dysfunction of blood coagulation(INR>2.0 or PT> 16s，APTT > 43s、TT > 21s，Fbg < 2g/L), having a tendency to bleed or undergoing thrombolysis or anticoagulant therapy; ascites with clinical symptoms, that is requiring therapeutic abdominal paracentesis or drainage or Child-Pugh score ≥2
* 17. Objective evidence of pulmonary fibrosis history, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug associated pneumonia, and severe lung function impairment in the past and at present
* 18. Urine routine showed that urine protein ≥++ or the urine protein in 24 hours>1.0 g
* 19. Patients who have been treated with potent CYP3A4 inhibitors (ketoconazole, itraconazole, voriconazole, ritonavir, clarithromycin, telithromycin, troleandomycin, erythromycin, cimetidine and so on) within 28 days before participating the study, or potent CYP3A4 inducers (dexamethasone, phenytoin, rifampin, rifabutin, carbamazepine, phenobarbitone and so on) within 12 days before participating the study
* 20. Pregnant or lactating women; fertile patients who are unwilling or unable to adopt effective contraceptives
* 21. Patients with mental sickness or the history of psychotropic drug abuse
* 22. Patients with severe infection (unable to control the infection effectively)
* 23. The treatment history affecting this program or its efficacy, such as stem cell transplantation, immune regulation (including PD-1 and other test regimens) recently (within half a year)
* 24. The researchers believe that any other factors unsuitable for entering into the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-07-18 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival | 24 months
  Time from start of treatment until the first documented event of symptomatic progression or death.

SECONDARY OUTCOMES:
Overall Survival | 36 months
  from start of treatment to death from any cause, or last known date of survival
large vascular invasion or extrahepatic metastasis (MVI/EHV) | 24 months
  The effect on large vascular invasion or extrahepatic metastasis (MVI/EHV)
Disease Control Rate (DCR) | 28 days
  the percentage of patients with advanced or metastatic cancer who have achieved complete response, partial response and stable disease
Objective Response Rate(ORR) | 28 days
  Proportion of patients with reduction in tumor burden of a predefined amount
biomarker | approximately 24 months
  decrease in tumor markers
quality of life | approximately 36 months
  The overall enjoyment of life.

CONTACTS AND LOCATIONS:
Overall Officials: Zujiang Yu, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China